CLINICAL TRIAL: NCT03281044
Title: Oral Frozen Fecal Microbiota Transplantation (FMT) Capsules for Depression: a Double-blind, Placebo-controlled, Randomized Parallel Group Study
Brief Title: Fecal Microbiota Transplantation in Depression
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Although not observed in our patients (4 enrolled), SAEs have been reported in other patients receiving the same product.
Sponsor: Psychiatric Hospital of the University of Basel (Other)
Responsible Party: Principal Investigator, André Schmidt, Research Group Leader, Psychiatric Hospital of the University of Basel
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2017-01050
Record Dates: First submitted 2017-09-04; First posted 2017-09-13 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FMT group (Experimental): Patient group receiving active FMT capsules
  Interventions: Drug: Fecal microbiota capsules
- Placebo group (Placebo Comparator): Patient group receiving placebo capsules
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Fecal microbiota capsules — Patients will receive FMT capsules DE containing the fecal microbiota drug substance within a gelatin capsule shell. The drug substance is fecal microbiota from a single donor.
  Arms: FMT group
Drug: Placebo oral capsule — The control condition is a placebo FMT capsule. The FMT placebo capsule is identical in appearance to active capsules, but does not contain human feces, the active pharmaceutical ingredient. Placebo capsules will contain an autoclaved solution of glycerol and saline, contained in an identical gelatin capsule as the active product, including the same enteric polymer coating
  Arms: Placebo group

SUMMARY:
The prevalence of psychiatric disorders such as major depression disorder (MDD) is increasing rapidly. Despite advancements in the development of therapeutics, current treatment options have not reached optimal efficacy.

Recent interest has been drawn towards the importance of the biochemical signalling between the gastrointestinal tract and the central nervous system also known as the "microbiome-gut-brain axis". The pathogenesis of gut microbiota in extra intestinal diseases was inspired by massive studies in germ free (GF) animals, which indicated that the gut microbiota plays a role in the normal regulation of behaviour that are relevant to mood, anxiety and stress. However, the exact mechanisms by which intestinal dysbiosis are involved in the development of psychiatric diseases are not completely clarified.

A new method to alter the composition of the gastrointestinal microbiota involves fecal microbiota transplantation (FMT). The goal of FMT is to introduce or restore a stable microbial community in the gut by transplanting intestinal microbiota from a healthy donor to the patient. FMT, as a microbiota-target therapy, is arguably very effective for curing recurrent Clostridium difficile infection and has good outcomes in other intestinal diseases. At the same time, applications in previously unexpected areas, including metabolic diseases, neuropsychiatric disorders, autoimmune diseases, allergic disorders, and tumors have shown health enhancing results. FMT has initially been conducted using colonoscopy. However, recent evidence has shown that treatment with frozen FMT capsules (to be taken orally) is also safe and beneficial in restoring the gut microbiota in patients with various diseases As FMT capsules may be an effective, pragmatical adjuvant therapy (in addition to standard treatment) for depression, this project is aimed at (1) investigating for the first time if single administration of FMT capsules ameliorates depressive symptoms in patients with moderate to severe MDD 4 weeks after treatment and (2) establishing the safety profile of encapsulated FMT in MDD. Furthermore, we will also test if (3) FMT capsules modulates immune signalling and inflammatory processes, (4) Hypothalamic-pituitary-adrenal (HPA) axis responses, (5) neurogenesis, (6) energy balance hormones, (7) gut microbiota composition and (8) brain perfusion, structure and activation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18, body mass index 20-30 kg/m²
* Able to provide signed and dated informed consent
* Patients with moderate to severe depression (as expressed by a Hamilton Depression Rating Scale (HAMD-17) > 17)
* Treatment as usual for depression
* In- and outpatients at the UPK Basel

Exclusion Criteria:

* Patients with mild MDD (HAMD-17 < 17)
* Comorbid psychiatric disturbances such as substance abuse disorder, bipolar disorder, schizophrenia, eating disorders.
* Current medical conditions such as acute infectious disease,
* Dietary restrictions (vegetarian, vegan, gluten-free, PEG/TPN feeding, and any kind of deviation from the UPK standard catering)
* Recent use of medications besides their anti-depressant medication (within 3 months, mainly antibiotics or probiotic consumption within last six weeks).
* Pregnancy (tested before both MRI scans using the AlereTM TestPack +Plus hCG Urine Test), breast-feeding
* Body Mass Index (BMI) > 30
* Current or recent use of antibiotics (within 3 months before inclusion)
* Anticipated antibiotic use in upcoming 4 weeks
* Inability to read and understand the participant's information and informed consent form
* Inability (e.g. dysphagia) to or unwilling to swallow capsules
* Active vomiting
* Known or suspected toxic megacolon and/or known small bowel ileus
* Major gastrointestinal surgery (e.g. significant bowel resection) within 3 months before enrolment. This does not include appendectomy or cholecystectomy.
* History of total colectomy or bariatric surgery.
* Concurrent intensive induction chemotherapy, radiation therapy or biological treatment for active malignancy. Patients on maintenance chemotherapy may be enrolled only after consultation with a medical monitor.
* Life expectancy < 6 months
* Patients with a history of severe anaphylactic or anaphylactoid food allergy
* Solid organ transplant recipients ≤ 90 days post-transplant or on active treatment for rejection
* Neuropenia (≤500 neutrophils/mL) or other severe immunosuppression. Anti-TNF will be permitted. Patients on monoclonal antibodies to B and T cells, glucocorticoids, antimetabolites (azathioprine, 6-mercaptopurine, methotrexate), calcineurin inhbitors (tacrolimus, cyclosporine) and mycophenolate mofetil may be enrolled only after consultation with the medical monitor.
* A condition that would jeopardize the safety or rights of the subject, would make it unlikely for the subject to complete the study, or would confound the results of the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2018-10-24 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-03-16 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms as measured with the Hamilton Rating Scale for Depression | Change from baseline score to follow-up measurements at 1, 2 and 8 months
  Efficacy measure

SECONDARY OUTCOMES:
Gut microbiota composition as assessed by 16-S-rRNA sequencing of stool samples | Change from baseline score to follow-up measurement after 1 month
  Efficacy measure
Cerebral blood flow (measured with arterial spin labeling, mL/100 g/min^10) | Change from baseline score to follow-up measurement after 1 month
  Efficacy measure
Brain structure (measured with structural magnetic resonance imaging to assess gray matter volume in mm^3, and diffusion tensor imaging to assess fractional anisotropy (dimensionless) and mean diffusivity (m2/s)) | Change from baseline score to follow-up measurement after 1 month
  Efficacy measure
Brain function (measured Blood-oxygen-level dependent contrast imaging) | Change from baseline score to follow-up measurement after 1 month
  Efficacy measure
HPA axis function (measured with salivary cortisol awakening responses). | Change from baseline score to follow-up measurement after 1 month
  Efficacy measure
Neurogenesis (measured with blood levels of BDNF). | Change from baseline score to follow-up measurement after 1 month
  Efficacy measure
Appetite-regulating hormones (measured with blood levels of ghrelin and leptin). | Change from baseline score to follow-up measurement after 1 month
  Efficacy measure
Immunoregulation and inflammation (measured with blood levels of macrophage migration inhibitory factor and interleukin 1 beta). | Change from baseline score to follow-up measurement after 1 month
  Efficacy measure
Cognition (measured with the Trail Making Test) | Change from baseline score to follow-up measurement after 1 month
  Efficacy measure
Physical activity (measured with a portable wristwatch). | Change from baseline score to follow-up measurement after 1 month
  Efficacy measure
Sleep quality (measured with 28-channel electroencephalography) | Change from baseline score to follow-up measurement after 1 month
  Efficacy measure

CONTACTS AND LOCATIONS:
Overall Officials: André Schmidt, Principal Investigator — University of Basel, Department of Psychiatry (UPK)
Locations (1):
- University Psychiatric Clinics (UPK), Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided